CLINICAL TRIAL: NCT03245840
Title: A Phase 3, Multicenter, Open-label Continuation Study With Budesonide Oral Suspension (BOS) for Adolescent and Adult Subjects With Eosinophilic Esophagitis (EoE)
Brief Title: Continuation Study With Budesonide Oral Suspension (BOS) for Adolescent and Adult Participants With Eosinophilic Esophagitis (EoE)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP621-303
Record Dates: First submitted 2017-08-08; First posted 2017-08-10 (Actual); Results first posted 2022-12-07 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2022-11

CONDITIONS: Eosinophilic Esophagitis (EoE)
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Budesonide Oral Suspension (Experimental): Participants received 10 milliliters (mL) of budesonide oral suspension at a concentration of 0.2 milligram per milliliter (mg/mL), twice daily, for up to 4 years 5 months.
  Interventions: Drug: Budesonide oral suspension

INTERVENTIONS:
Drug: Budesonide oral suspension — BOS 10 mL twice daily.

SUMMARY:
This is a continuation study of Budesonide Oral Suspension (BOS) in adults and adolescents with Eosinophilic Esophagitis (EoE) who have completed participation in the SHP621-302 extension study. The purpose of this study is to see if BOS is safe and well tolerated over the long-term in adolescents and adults with EoE.

ELIGIBILITY:
Inclusion Criteria:

* Participant completed the SHP621-302 (NCT02736409) extension study and is considered by the investigator to potentially benefit from continued BOS investigational treatment.
* Participant is able to provide written informed consent (participant, parent or legal guardian and, as appropriate, participant assent) to participate in the study before completing any study-related procedures.
* Females of childbearing potential must agree to continue acceptable birth control measures (example (e.g.): abstinence, surgically sterile male partner, stable oral contraceptives, or double-barrier methods) throughout study participation.
* Participant is willing and has an understanding and ability to fully comply with study procedures and restrictions as defined in protocol.

Exclusion Criteria:

* Participant has changes in medications or diet during the SHP621-302 (NCT02736409) study that could affect participation in this continuation study.
* Participant anticipates using swallowed topical corticosteroid for EoE or systemic corticosteroid for any condition during the treatment period; any temporary use (less than or equal to [≤] 7 days) or initiation of new steroid treatment during the study should be documented and discussed with the medical monitor prospectively but should be avoided within 4 weeks of the scheduled esophagogastroduodenoscopy (EGDs).
* Participant anticipates use of Cytochrome P450 3A4 inhibitors (e.g., ketoconazole, grapefruit juice) during the continuation study.
* Participant has an appearance at the EGD at the final treatment evaluation visit of SHP621-302 (NCT02736409) (Visit 8) of an esophageal stricture (high grade), as defined by the presence of a lesion that does not allow passage of a diagnostic adult upper endoscope (e.g., with an insertion tube diameter of greater than (>) 9 millimeter [mm]).
* Participant has presence of esophageal varices at the EGD at the final treatment evaluation visit (Visit 8) of the SHP621-302 (NCT02736409) study.
* Participant has any current disease of the gastrointestinal tract, aside from EoE, including eosinophilic gastritis, enteritis, colitis, or proctitis, inflammatory bowel disease, or celiac disease.
* Participant has other diseases causing or associated with esophageal eosinophilia, including hypereosinophilic syndrome, collagen vascular disease, vasculitis, achalasia, or parasitic infection.
* Participant has oropharyngeal or esophageal candidiasis that failed to respond to previous treatment. Diagnosis with oropharyngeal or esophageal candidiasis at or since the final treatment evaluation visit (Visit 8) of the SHP621-302 (NCT02736409) study is not an exclusion as long as the participant is expected to respond to treatment.
* Participant has a potentially serious acute or chronic infection or immunodeficiency condition, including tuberculosis, fungal, bacterial, viral/parasite infection, ocular herpes simplex, or chicken pox/measles.
* Participant has upper gastrointestinal bleeding identified at the EGD at the final treatment evaluation visit (Visit 8) of the SHP621-302 (NCT02736409) study.
* Participant has evidence of active infection with Helicobacter pylori.
* Participant has evidence of unstable asthma.
* Participant is female and pregnant or nursing.
* Participant has a history of intolerance, hypersensitivity, or idiosyncratic reaction to budesonide (or any other corticosteroids), or to any other ingredients of the study medication.
* Participant has a history or high risk of noncompliance with treatment or regular clinic visits.

Ages: 11 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 133 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (45):
- United States (45):
  - Children's Hospital, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Del Sol Research Management, Tucson, Arizona
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Rady Children's Hospital San Diego, San Diego, California
  - Colorado Children's Hospital, Aurora, Colorado
  - Asthma and Allergy Associates PC, Colorado Springs, Colorado
  - Rocky Mountain Pediatric Gastroenterology, Denver, Colorado
  - Connecticut Clinical Research Foundation, Bristol, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Connecticut GI, Hartford, Connecticut
  - Nature Coast Clinical Research LLC, Inverness, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Childrens Center For Digestive Healthcare, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Grand Teton Research Group, Idaho Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - Gastroenterology of Southern Indiana, New Albany, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Indiana University, Louisville, Kentucky
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Clinical Trials Management LLC, Metairie, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital, Chestnut Hill, Massachusetts
  - Minnesota Gastroenterology PA, Plymouth, Minnesota
  - Mount Sinai Hospital, Icahn School of Medicine, Astoria, New York
  - Long Island Gastrointestinal Research Group LLP, Great Neck, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Gastrointestinal and Liver Diseases Consultants PC, Dayton, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - Digestive Disease Specialists, Inc., Oklahoma City, Oklahoma
  - Greenville Hospital, Greenville, South Carolina
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Endoscopy and Research Center, Houston, Texas
  - Advanced Research Institute, Ogden, Utah
  - Primary Children's Hospital, University of Utah, Salt Lake City, Utah
  - Emeritas Research Group, Lansdowne Town Center, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as the data are subject to contractual (or consent) provisions that prohibit transfer to third parties.

REFERENCES:
- [Derived] Dellon ES, Katzka DA, Mukkada VA, Collins MH, Falk GW, Richmond CA, Terreri B, Thakur M, Boules M, Goodwin B, Hirano I. Long-term Safety and Efficacy of Budesonide Oral Suspension for Eosinophilic Esophagitis: A 4-Year, Phase 3, Open-Label Study. Clin Gastroenterol Hepatol. 2025 Nov;23(12):2155-2166.e5. doi: 10.1016/j.cgh.2024.12.024. Epub 2025 Feb 13. PMID 39954913
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fd84db2bf003ab47062

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 44 active sites in North America from 05 October 2017 (first participant enrolled) to 26 April 2022 (last participant completed).
Pre-assignment Details: A total of 174 participants completed the study SHP621-302 (NCT02736409), of which 133 consented to participate and were enrolled in this long-term safety and efficacy study (SHP621-303). A total of 131 participants were treated in this study. This study was terminated as per sponsor's decision.
Groups:
- BOS-BOS: Participants who were randomized to budesonide oral suspension (BOS) and placebo (PBO) in Study SHP621-301 (NCT02605837) and to BOS in Study SHP621-302 (NCT02736409), were enrolled in Study SHP621-303 to receive 10 milliliters (mL) of BOS at a concentration of 0.2 milligram per milliliter (mg/mL), twice daily, for up to 4 years 5 months.
- PBO-BOS: Participants who were randomized to and fully responded to BOS treatment in Study SHP621-301 (NCT02605837), were randomized to PBO in Study SHP621-302 (NCT02736409) and enrolled in Study SHP621-303 to receive 10 mL of BOS at a concentration of 0.2 mg/mL, twice daily, for up to 4 years 5 months.
Period: Overall Study
Arm/Group | BOS-BOS | PBO-BOS
Started | 122 | 11
Treated | 121 | 10
Completed | 0 | 0
Not Completed | 122 | 11
Not completed — Adverse Event | 6 | 0
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 31 | 1
Not completed — Withdrawal by Parent/Guardian | 2 | 0
Not completed — Physician Decision | 4 | 1
Not completed — Study Terminated by Sponsor | 56 | 6
Not completed — Site Terminated by Sponsor | 4 | 0
Not completed — Lost to Follow-up | 12 | 2
Not completed — Pregnancy | 2 | 0
Not completed — Non-Compliance with Study Drug | 2 | 0
Not completed — Not treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAS) consisted of all participants who received at least 1 dose of BOS.
Groups:
- BOS-BOS: Participants who were randomized to BOS and PBO in Study SHP621-301 (NCT02605837) and to BOS in Study SHP621-302 (NCT02736409), were enrolled in Study SHP621-303 to receive 10 mL of BOS at a concentration of 0.2 mg/mL, twice daily, for up to 4 years 5 months.
- Total: Total of all reporting groups
Arm/Group | BOS-BOS | PBO-BOS | Total
Number analyzed (Participants) | 121 | 10 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (12.65) | 40.2 (9.97) | 34.4 (12.55)
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 22 | 0 | 22
  18 or more years | 99 | 10 | 109
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 2 | 49
  Male | 74 | 8 | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 117 | 10 | 127
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 0 | 4
  White | 109 | 10 | 119
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. A Serious Adverse Event (SAE) was any untoward medical occurrence (whether considered to be related to investigational product or not) that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital abnormality/birth defect, and is an important medical event. Both serious and Non-serious TEAEs were reported in this outcome measure. TEAEs were defined as AEs with a start date on or after the first dose of investigational product or a start date before the date of the first dose of investigational product that increased in severity or after the date of the first dose.
Time Frame: From start of study drug administration up to End of study (EOS) (Up to Month 53)
Population: The safety set consisted of all participants who received at least 1 dose of BOS.
Measure: Count of Participants; unit: Participants
Arm/Group | BOS-BOS | PBO-BOS
Number analyzed (Participants) | 121 | 10
Participants
  TEAEs | 93 | 7
  Serious TEAEs | 11 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Physical Examination Findings
Description: Number of participants with clinically significant physical examination findings were reported. Clinical significance was determined by investigator.
Time Frame: From start of study drug administration up to EOS (Up to Month 53)
Population: The safety set consisted of all participants who received at least 1 dose of BOS.
Measure: Count of Participants; unit: Participants
Arm/Group | BOS-BOS | PBO-BOS
Number analyzed (Participants) | 121 | 10
Participants
  Moon Face | 0 | 0
  Acne | 2 | 0
  Hirsutism | 0 | 0
  Mood swings | 0 | 0
  Insomnia | 0 | 0
  Depression | 1 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Participants were assessed by investigator for any clinically significant changes in vital parameters like temperature, systolic and diastolic blood pressure, pulse, respiratory rate, BMI, and weight. Vital signs were assessed after the participant had been in a supine position for at least 5 minutes immediately prior to the assessment. The criteria for clinically significant change was as per the investigators discretion.
Time Frame: From start of study drug administration up to EOS (Up to Month 53)
Population: The safety set consisted of all participants who received at least 1 dose of BOS.
Measure: Count of Participants; unit: Participants
Arm/Group | BOS-BOS | PBO-BOS
Number analyzed (Participants) | 121 | 10
Participants | 0 | 0

4. Primary Outcome: Change From Baseline in Bone Mineral Density (BMD) For Adolescents Assessed by Dual-Energy X-ray Absorptiometry (DXA) Scan at Month 12
Description: The sites for DXA measurement were the lumbar spine at lumbar vertebrae 1 to 4 (L1-L4) and whole body. DXA scans for determination of BMD and body composition was performed in participants aged 11-17 years. Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. In this study, the BMD Z-score is considered abnormal when the z-score is less than (<) -2, suggesting a worse outcome (i.e., osteoporosis). Change from baseline in BMD for adolescents assessed by DXA Scan at Month 12 was reported.
Time Frame: Baseline, Month 12
Population: The safety set consisted of all participants who received at least 1 dose of BOS. Here, overall number of participants analyzed signified participants who were evaluable for this outcome measure and number analyzed signifies participants who were evaluable for given categories. DXA was performed for participants aged 11-17 years only and no participants of this age range were present in PBO-BOS group.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | BOS-BOS
Number analyzed (Participants) | 18
Z-score
  Baseline Lumbar Spine (L1- L4) | -0.525 (1.0583)
  Change at Month 12 Lumbar Spine (L1- L4): number analyzed (Participants) | 8
  Change at Month 12 Lumbar Spine (L1- L4) | 0.315 (0.3618)
  Baseline Whole Body | -0.565 (0.9464)
  Change at Month 12 Whole Body: number analyzed (Participants) | 8
  Change at Month 12 Whole Body | 0.250 (0.2599)

5. Primary Outcome: Change From Baseline in BMD For Adolescents Assessed by DXA Scan at Month 24
Description: The sites for DXA measurement were the lumbar spine at lumbar vertebrae 1 to 4 (L1-L4) and whole body. DXA scans for determination of BMD and body composition was performed in participants aged 11-17 years. Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. In this study, the BMD Z-score is considered abnormal when the z-score is <-2, suggesting a worse outcome (i.e., osteoporosis) and vice versa. Change from baseline in BMD for adolescents assessed by DXA Scan at Month 24 was reported.
Time Frame: Baseline, Month 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | BOS-BOS
Number analyzed (Participants) | 18
Z-score
  Baseline Lumbar Spine (L1- L4) | -0.525 (1.0583)
  Change at Month 24 Lumbar Spine (L1- L4): number analyzed (Participants) | 12
  Change at Month 24 Lumbar Spine (L1- L4) | 0.445 (0.7312)
  Baseline Whole Body | -0.565 (0.9464)
  Change at Month 24 Whole Body: number analyzed (Participants) | 11
  Change at Month 24 Whole Body | 0.092 (0.5326)

6. Primary Outcome: Change From Baseline in BMD For Adolescents Assessed by DXA Scan at Month 36
Description: The sites for DXA measurement were the lumbar spine at lumbar vertebrae 1 to 4 (L1-L4) and whole body. DXA scans for determination of BMD and body composition was performed in participants aged 11-17 years. Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. In this study, the BMD Z-score is considered abnormal when the z-score is < -2, suggesting a worse outcome (i.e., osteoporosis) and vice versa. Change from baseline in BMD for adolescents assessed by DXA Scan at Month 36 was reported.
Time Frame: Baseline, Month 36
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | BOS-BOS
Number analyzed (Participants) | 18
Z-score
  Baseline Lumbar Spine (L1- L4) | -0.525 (1.0583)
  Change at Month 36 Lumbar Spine (L1- L4): number analyzed (Participants) | 4
  Change at Month 36 Lumbar Spine (L1- L4) | 0.603 (0.9089)
  Baseline Whole Body | -0.565 (0.9464)
  Change at Month 36 Whole Body: number analyzed (Participants) | 4
  Change at Month 36 Whole Body | 0.870 (0.6447)

7. Primary Outcome: Change From Baseline in BMD For Adolescents Assessed by DXA Scan at Month 48
Description: The sites for DXA measurement were the lumbar spine at lumbar vertebrae 1 to 4 (L1-L4) and whole body. DXA scans for determination of BMD and body composition was performed in participants aged 11-17 years. Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. In this study, the BMD Z-score is considered abnormal when the z-score is < -2, suggesting a worse outcome (i.e., osteoporosis) and vice versa. Change from baseline in BMD for adolescents assessed by DXA Scan at Month 48 was reported.
Time Frame: Baseline, Month 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | BOS-BOS
Number analyzed (Participants) | 18
Z-score
  Baseline Lumbar Spine (L1- L4) | -0.525 (1.0583)
  Change at Month 48 Lumbar Spine (L1- L4): number analyzed (Participants) | 3
  Change at Month 48 Lumbar Spine (L1- L4) | 0.657 (0.4813)
  Baseline Whole Body | -0.565 (0.9464)
  Change at Month 48 Whole Body: number analyzed (Participants) | 3
  Change at Month 48 Whole Body | 0.817 (0.4521)

8. Primary Outcome: Change From Baseline in BMD For Adolescents Assessed by DXA Scan at EOS (Up to Month 53)
Description: The sites for DXA measurement were the lumbar spine at lumbar vertebrae 1 to 4 (L1-L4) and whole body. DXA scans for determination of BMD and body composition was performed in participants aged 11-17 years. Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. In this study, the BMD Z-score is considered abnormal when the z-score is < -2, suggesting a worse outcome (i.e., osteoporosis) and vice versa. Change from baseline in BMD for adolescents assessed by DXA Scan at EOS (up to Month 53) was reported.
Time Frame: Baseline, EOS (Up to Month 53)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | BOS-BOS
Number analyzed (Participants) | 18
Z-score
  Baseline Lumbar Spine (L1- L4) | -0.525 (1.0583)
  Change at EOS (Up to Month 53) Lumbar Spine (L1- L4): number analyzed (Participants) | 13
  Change at EOS (Up to Month 53) Lumbar Spine (L1- L4) | 0.482 (0.6539)
  Baseline Whole Body | -0.565 (0.9464)
  Change at EOS (Up to Month 53) Whole Body: number analyzed (Participants) | 13
  Change at EOS (Up to Month 53) Whole Body | 0.350 (0.7541)

9. Primary Outcome: Change From Baseline in Cortisol Level After Adrenocorticotropic Hormone (ACTH) Stimulation at Month 12
Description: ACTH testing was a standard procedure to measure the levels of cortisol in the blood following the injection of a synthetic form of ACTH (250 microgram [mcg]). The type of synthetic and route of administration was per investigator discretion. The change from baseline in cortisol levels was calculated at Month 12 and reported in this outcome measure.
Time Frame: Baseline, Month 12
Population: The safety set consisted of all participants who received at least 1 dose of BOS. Here, overall number of participants analyzed signified participants who were evaluable for this outcome measure and number analyzed signifies participants who were evaluable for given categories.
Measure: Mean (Standard Deviation); unit: micrograms per deciliter (mcg/dL)
Arm/Group | BOS-BOS | PBO-BOS
Number analyzed (Participants) | 118 | 10
micrograms per deciliter (mcg/dL)
  Baseline | 10.49 (5.508) | 13.15 (7.188)
  Change At Month 12: number analyzed (Participants) | 84 | 6
  Change At Month 12 | 0.06 (6.215) | 6.77 (8.835)

10. Primary Outcome: Change From Baseline in Cortisol Level After ACTH Stimulation at Month 24
Description: ACTH testing was a standard procedure to measure the levels of cortisol in the blood following the injection of a synthetic form of ACTH (250 microgram [mcg]). The type of synthetic and route of administration was per investigator discretion. The change from baseline in cortisol levels was calculated at Month 24 and reported in this outcome measure.
Time Frame: Baseline, Month 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | BOS-BOS | PBO-BOS
Number analyzed (Participants) | 118 | 10
mcg/dL
  Baseline | 10.49 (5.508) | 13.15 (7.188)
  Change At Month 24: number analyzed (Participants) | 77 | 6
  Change At Month 24 | 0.81 (6.127) | -2.58 (3.727)

11. Primary Outcome: Change From Baseline in Cortisol Level After ACTH Stimulation at Month 36
Description: ACTH testing was a standard procedure to measure the levels of cortisol in the blood following the injection of a synthetic form of ACTH (250 microgram [mcg]). The type of synthetic and route of administration was per investigator discretion. The change from baseline in cortisol levels was calculated at Month 36 and reported in this outcome measure.
Time Frame: Baseline, Month 36
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | BOS-BOS | PBO-BOS
Number analyzed (Participants) | 118 | 10
mcg/dL
  Baseline | 10.49 (5.508) | 13.15 (7.188)
  Change At Month 36: number analyzed (Participants) | 66 | 6
  Change At Month 36 | 0.70 (5.773) | -1.63 (3.845)

12. Primary Outcome: Change From Baseline in Cortisol Level After ACTH Stimulation at Month 48
Description: ACTH testing was a standard procedure to measure the levels of cortisol in the blood following the injection of a synthetic form of ACTH (250 microgram [mcg]). The type of synthetic and route of administration was per investigator discretion. The change from baseline in cortisol levels was calculated at Month 48 and reported in this outcome measure.
Time Frame: Baseline, Month 48
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | BOS-BOS | PBO-BOS
Number analyzed (Participants) | 118 | 10
mcg/dL
  Baseline | 10.49 (5.508) | 13.15 (7.188)
  Change At Month 48: number analyzed (Participants) | 26 | 4
  Change At Month 48 | 2.02 (4.759) | 0.20 (5.170)

13. Primary Outcome: Change From Baseline in Cortisol Level After ACTH Stimulation at EOS (Up to Month 53)
Description: ACTH testing was a standard procedure to measure the levels of cortisol in the blood following the injection of a synthetic form of ACTH (250 microgram [mcg]). The type of synthetic and route of administration was per investigator discretion. The change from baseline in cortisol levels was calculated at EOS (up to Month 53) and reported in this outcome measure.
Time Frame: Baseline, EOS (Up to Month 53)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | BOS-BOS | PBO-BOS
Number analyzed (Participants) | 118 | 10
mcg/dL
  Baseline | 10.49 (5.508) | 13.15 (7.188)
  Change at EOS (Up to Month 53): number analyzed (Participants) | 83 | 7
  Change at EOS (Up to Month 53) | 0.96 (5.362) | 1.06 (6.138)

14. Primary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Assessments
Description: Clinical laboratory parameters included hematology, chemistry, urinalysis; urine pregnancy test. Number of participants with potential clinically significant changes in laboratory parameters which were deemed clinically meaningful by the investigator were reported.
Time Frame: From start of study drug administration up to EOS (Up to Month 53)
Population: The safety set consisted of all participants who received at least 1 dose of BOS.
Measure: Count of Participants; unit: Participants
Arm/Group | BOS-BOS | PBO-BOS
Number analyzed (Participants) | 121 | 10
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to EOS (Up to Month 53)
Description: The safety set consisted of all participants who received at least 1 dose of BOS.
Arm/Group | BOS-BOS | PBO-BOS
All-Cause Mortality (participants affected / at risk) | 2/121 | 0/10
Serious Adverse Events (participants affected / at risk) | 11/121 | 0/10
Other Adverse Events (participants affected / at risk) | 90/121 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BOS-BOS (N=121) | PBO-BOS (N=10)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BOS-BOS (N=121) | PBO-BOS (N=10)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 8 (8) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 1 (1)
Oesophageal food impaction (Gastrointestinal disorders) | 5 (9) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 2 (4) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Corona virus infection (Infections and infestations) | 10 (10) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 7 (7) | 0 (0)
Nasopharyngitis (Infections and infestations) | 8 (9) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 4 (5) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 10 (11) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ACTH stimulation test abnormal (Investigations) | 14 (16) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1)
Depression (Psychiatric disorders) | 10 (12) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Obsessive-compulsive disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Hypertension (Vascular disorders) | 7 (7) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was discontinued prematurely as per sponsor's decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT03245840/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT03245840/SAP_001.pdf